CLINICAL TRIAL: NCT04909606
Title: Evaluation of a Nurse-led Program for the Prevention of Complications of Long-term Corticosteroid Therapy
Acronym: COCORTICO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 29BRC20.0119
Record Dates: First submitted 2021-04-23; First posted 2021-06-02 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Long Term Corticosteroid Therapy
Keywords: Nurse-led program; Prevention; Corticosteroids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nurse-led prevention program (Experimental): Patients will receive a general summary sheet of preventive measures associated with long term corticosteroids therapy (no individual assessment) in addition to the usual care provided by their physician
  Interventions: Other: nurse-led prevention program
- Standard of care (Active Comparator): Subjects randomized to the nurse-led prevention program group will be evaluated by the dedicated nurse within 2 weeks following randomization (individual assessment)
  Interventions: Other: Current care

INTERVENTIONS:
Other: nurse-led prevention program — Subjects randomized to the nurse-led prevention program group will be evaluated by the dedicated nurse within 2 weeks following randomization (individual assessment)
  The nurse-led prevention program will include:
  1. A video explaining corticosteroids related adverse events and adequate preventive measures
  2. An individual interview with the trained nurse
  3. A consultation with a dietetician
  4. An individual sheet summarizing appropriate non-pharmacological preventive measures for the participant
  5. An individual sheet summarizing appropriate pharmacological preventive measures for the referent physician
  6. Phone calls at week-12, week-24 and week-36 to ensure the appropriate implementation of preventive measures
  Arms: Nurse-led prevention program
Other: Current care — Subjects randomized to the standard of care group will receive a general summary sheet of preventive measures associated with long term corticosteroids therapy (no individual assessment) in addition to the usual care provided by their physician
  Arms: Standard of care

SUMMARY:
Long term corticosteroid therapy concerns 0.5 to 1% of the population and about 2.5% of elderly subjects. It is currently used as a cornerstone therapy in a wide variety of clinical contexts. The central problematic of prolonged corticosteroid therapy is the burden of adverse events associated with its long term use, including bone, metabolic and infectious complications.

The management of patients for whom the prescription of long term corticosteroid therapy is indicated should include an evaluation of the individual risk and implementation of the appropriate preventive measures. Such an approach should particularly include cortisonic osteoporosis prevention, infectious prevention including vaccination, prevention of adrenal insufficiency, promotion of physical activity, as well as dietary management.

In France, nurse-led prevention programs are highly developed for patients initiating immunosuppressive targeted therapies. Conversely, there are no dedicated nurse-led programs for patients starting prolonged corticosteroid therapy, for several historical and economical reasons.

The implementation of such programs is likely to be beneficial at different levels, including the reduction of the number of adverse events and improvement of health-related quality of life.

The main objective of the study is to determine the long-term benefit of a nurse-led prevention program among patients starting long-term corticosteroids therapy, compared to routine care.

DETAILED DESCRIPTION:
It is a PROBE (Prospective Randomized Open trial with a Blind Evaluation) study, in which the primary endpoint will be assessed at week-52 by an independent physician blinded to the participant's allocation group.

The target population is adult patients initiating a first sequence of long term corticosteroid therapy, to the exception of onco-hematological indications, severe chronic renal failure and organ transplant.

Patients in both groups will have baseline and week-52 standardized visits including clinical evaluation, routine biology, dual-energy X-ray absorptiometry and quality of life assessment (SF-36). Corticosteroid consumption will be collected throughout the study using a dedicated notebook. At the week-52 visit, the burden of adverse events related to the use of corticosteroids will be assessed through the glucocorticoid toxicity index (GTI), completed by the blinded physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older
* Initiation of corticosteroids within 30 days prior to inclusion
* Estimated cumulative dosage of corticosteroids ≥ 2000 mg
* Affiliated member of the social security system

Exclusion Criteria:

* Patients unable to give consent or unable to understand the protocol
* A patient who is not 'or is no longer' able to communicate remotely by telephone could not 'or no longer' be included in the study.
* Patients under guardianship
* Previous exposure to long-term corticosteroids
* Prescription of corticosteroids for the management of malignant neoplasms
* Severe chronic renal failure with clearance of creatinine < 30 ml/min.
* History of organ transplantation
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Determine the ability of a prevention program to reduce the burden of adverse events attributable to corticosteroid therapy | 12 months
  Glucocorticoid Toxicity Index Raw Score

SECONDARY OUTCOMES:
occurrence of at least one clinically significant complication of steroid therapy | 12 months
  binary criterion derived from the glucocorticoid toxicity index.
Following of the quality of life | 12 months
  The Short Form 36 (SF36) is used to evaluate the quality of life.
The occurrence of different categories of complications of long-term corticosteroid therapy | 12 months
  Complication categories defined by the glucocorticoid toxicity index
Application of preventive drug measures | 12 months
  Immunization record
Cumulative glucocorticoid dosage actually received | 12 months
  Cumulative dosage estimated at week 52 using a compliance logbook completed by the patient

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU Brest, Brest
  - CH La Rochelle, La Rochelle
  - CH Le Mans, Le Mans
  - CH Le Puy en Velay, Le Puy-en-Velay
  - CH de Morlaix, Morlaix

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Derived] Nicol S, Trin K, Simon LA, Nowak E, Duval O, Martin C, Abdelouahad S, Lengagne S, Chinchilla V, Gilet V, Briantais A, Saraux A, Cornec D, De Moreuil C, Tanguy ML, Guellec D. Evaluation of a nurse-led program for the prevention of complications of long-term glucocorticoids (COCORTICO): study protocol for a randomized trial. Trials. 2025 Nov 17;26(1):510. doi: 10.1186/s13063-025-09236-4. PMID 41250159